CLINICAL TRIAL: NCT02285166
Title: Specified Drug-use Survey of Lotriga Granular Capsules: OCEAN3 (Outcome Prevention on Cardiovascular Events by Antihyperlipidemic Therapy With N3-fatty Acid in Japan)
Brief Title: Specified Drug-use Survey of the Granular Capsule Formulation of Omega-3 Fatty Acid Ethyl Esters: OCEAN3
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 142-012; JapicCTI-142680 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-07

CONDITIONS: Hyperlipidemia
Keywords: Pharmacological therapy
MeSH Terms: conditions — Hyperlipidemias | interventions — Omacor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ever User of Omega-3 fatty acid ethyl esters 2 g: The usual adult dosage for oral use was 2 g of omega-3 fatty acid ethyl esters administered once daily or twice daily immediately after meals for treatment of hyperlipidemia. Participants received both interventions and standard antihyperlipidemic therapy as part of routine medical care.
  Interventions: Drug: Omega-3 fatty acid ethyl esters
- Never User of Omega-3 fatty acid ethyl esters 2 g: Participants received standard antihyperlipidemic therapy without omega-3 fatty acid ethyl esters 2 g as part of routine medical care.
  Interventions: Drug: Standard antihyperlipidemic therapy other than administration of omega-3 fatty acid ethyl esters (Lotriga).

INTERVENTIONS:
Drug: Omega-3 fatty acid ethyl esters — Omega-3 fatty acid ethyl esters granular capsules
  Other Names: Lotriga granular capsules
  Groups: Ever User of Omega-3 fatty acid ethyl esters 2 g
Drug: Standard antihyperlipidemic therapy other than administration of omega-3 fatty acid ethyl esters (Lotriga).
  Groups: Never User of Omega-3 fatty acid ethyl esters 2 g

SUMMARY:
The purpose of this survey is to determine the incidence rate of cardiovascular (CV) events associated with long-term treatment with and without omega-3 fatty acid ethyl esters (Lotriga Granular Capsules) in high-risk hyperlipidemic patients treated by statin in daily medical practice.

DETAILED DESCRIPTION:
This survey is planned to determine the incidence rate of cardiovascular (CV) events associated with long-term treatment with omega-3 fatty acid ethyl esters (Lotriga Granular Capsules) in high-risk hyperlipidemic patients treated by statin in daily medical practice.

The incidence rate of CV events in the participants who are treated by the standard anti-hyperlipidemic therapies other than omega-3 fatty acid ethyl esters is investigated in this survey so as to compare the events rates between two participant groups just for information.

For adults, 2 g of omega-3 fatty acid ethyl esters is usually administered orally once daily immediately after meals. However, the dose can be increased up to twice daily (to a dose of 2 g) depending on participant's triglyceride (TG) level.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all of the following criteria will be included in the survey:

1. Patients with hyperlipidemia on statin therapy
2. Outpatients
3. Male participants aged ≥ 50 years and female participants aged ≥ 60 years
4. Participants with fasting TG level ≥ 150 mg/dL (within 3 months prior to the start of the observation period)
5. Participants who have at least two of the following risk factors:

   * Hypertension
   * Type 2 diabetes mellitus
   * Chronic kidney disease
   * Prior history of myocardial infarction or angina pectoris
   * Prior history of cerebral infarction
   * Peripheral arterial disease

Exclusion Criteria:

-Participants who meet any of the following criteria will be excluded from the survey:

1. Participants who have experienced coronary artery disease within 1 month prior to the start of the observation period
2. Participants who have experienced cerebrovascular disease within 1 month prior to the start of the observation period
3. Participants who have undergone heart surgery or revascularization surgery (including coronary artery intervention and peripheral arterial intervention) within 1 month prior to the start of the observation period
4. Participants who plan to undergo heart surgery or revascularization surgery (including coronary artery intervention and peripheral arterial intervention)
5. Patients with malignant tumors currently under treatment
6. Participants who have received eicosapentaenoic acid (hereinafter, EPA) products within 1 month prior to the start of the observation period, or participants who plan to receive treatment with EPA products after the start of the observation period
7. Patients with hemorrhage (e.g., hemophilia, capillary fragility, gastrointestinal ulcer, urinary tract hemorrhage, hemoptysis, or vitreous hemorrhage)
8. Participants with prior history of hypersensitivity to any ingredients in omega-3 fatty acid ethyl esters (omega-3 fatty acid ethyl esters-treated participants only)
9. Participants with prior history of treatment with omega-3 fatty acid ethyl esters

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hyperlipidemia
Sampling Method: Non-Probability Sample
Enrollment: 15330 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Teramoto T, Ogawa H, Ueshima H, Okada Y, Haze K, Matsui S, Fujikawa K, Hashimoto T, Sakui S, Nishimura K, Kajita M, Horimoto A, Fernandez J. Effect of omega-3 fatty acids on cardiovascular events in high-risk patients with hypertriglyceridemia in Japan: a 3-year post-marketing surveillance study (OCEAN3 survey). Expert Opin Drug Saf. 2023 Jan;22(1):81-90. doi: 10.1080/14740338.2022.2094914. Epub 2022 Jul 8. PMID 35772177
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60164db2bf003ab490aa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 1076 investigative sites in Japan, from 21 October 2014 to 14 July 2020.
Pre-assignment Details: High-risk hyperlipidemic patients treated by statin in daily medical practice were enrolled. Participants received standard antihyperlipidemic therapy with or without intervention of omega-3 fatty acid ethyl esters as part of a routine medical care. Reported groups were combined because group assignment (With/Without intervention) was conducted after completion of data collection in this observational study and data collection for each group was not planned on the protocol of this study.
Groups:
- Overall: Participants received standard antihyperlipidemic therapy with or without intervention of omega-3 fatty acid ethyl esters by the end of surveillance as part of a routine medical care.
Period: Overall Study
Arm/Group | Overall
Started | 15330
Completed | 14364
Not Completed | 966
Not completed — Case Report Forms Uncollected | 564
Not completed — Protocol Deviation | 402

BASELINE CHARACTERISTICS:
Population: Efficacy Analysis Set, The efficacy analysis set was defined as all participants who completed the survey. Reported groups were combined in this section because group assignment (groups with or without intervention of omega-3 fatty acid ethyl esters) was conducted after completion of data collection (collection of Case Report Form) in this observational study and collection of data for each group during this study was not planned on the protocol of this study.
Arm/Group | Overall
Number analyzed (Participants) | 14364
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.8 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6499
  Male | 7865
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 14364
Number of Risk Factors [Count of Participants; unit: Participants] — Number of participants who had 2 or more risk factors at baseline was reported. Risk factors were categorized as follows; High blood pressure, Type 2 diabetes, Chronic kidney disease, History of myocardial infarction or angina, History of cerebral infarction, Peripheral artery disease.
  Participants
    2 | 9749
    3 | 3532
    4 | 919
    5 | 150
    6 | 14
Onset Time of Myocardial Infarction before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced myocardial infarction before study start as past medical history.
  Participants
    number analyzed (Participants) | 1261
    Less than 1 year | 102
    More than 1 year ago | 1159
Frequency of Onset of Myocardial Infarction before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced myocardial infarction before study start as past medical history.
  Participants
    number analyzed (Participants) | 1261
    Once | 1202
    Twice | 47
    More than 3 times | 12
Onset Time of Cerebral Infarction before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced cerebral infarction before study start as past medical history.
  Participants
    number analyzed (Participants) | 2224
    Less than 1 year | 199
    More than 1 year ago | 2025
Frequency of Onset of Cerebral Infarction before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced cerebral infarction before study start as past medical history.
  Participants
    number analyzed (Participants) | 2224
    Once | 2086
    Twice | 93
    More than 3 times | 45
Number of Participants Who Underwent Coronary Revascularization [Count of Participants; unit: Participants]
  Not received | 12463
  Received | 1901
History of Peripheral Arterial Intervention [Count of Participants; unit: Participants]
  Not received | 14207
  Received | 157
BMI [Mean (Standard Deviation); unit: Kilogram (kg)/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  Kilogram (kg)/meter (m)^2
    number analyzed (Participants) | 12982
    (all) | 25.39 (3.782)
Smoking Classification [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 13866
    Never Smoked | 7574
    Current Smoker | 1825
    Ex-Smoker | 4467
Drinking Habits [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 13890
    Drink 5 days or more per week | 3645
    Drink less than 5 days per week or not drink | 10245
Frequency of Hospital Visit [Count of Participants; unit: Participants]
  More than twice a month | 1410
  Around once a month | 9191
  Once or twice every 3 months | 3596
  Less than once or twice every 3 months | 167
Frequency of Fish Consumption [Count of Participants; unit: Participants]
  Almost everyday | 1234
  Around once every other day | 4272
  Around once or twice a week | 6838
  Rarely eat | 984
  Data not available | 1036
History and Complications of Cerebro-cardiovascular Disorder [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 14240
    Presence | 11947
    Absence | 2293
Onset Time of Cerebral Hemorrhage before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced cerebral hemorrhage before study start as past medical history.
  Participants
    number analyzed (Participants) | 167
    Less than 1 year | 8
    More than 1 year ago | 159
Frequency of Onset of Cerebral Hemorrhage before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced cerebral hemorrhage before study start as past medical history.
  Participants
    number analyzed (Participants) | 167
    Once | 153
    Twice | 10
    More than 3 times | 1
    Data not available | 3
Onset Time of Subarachnoid Hemorrhage before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced subarachnoid hemorrhage before study start as past medical history.
  Participants
    number analyzed (Participants) | 44
    Less than 1 year | 3
    More than 1 year ago | 41
Frequency of Onset of Subarachnoid Hemorrhage before Study Start [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis who experienced subarachnoid hemorrhage before study start as past medical history.
  Participants
    number analyzed (Participants) | 44
    Once | 44
    Twice | 0
    More than 3 times | 0
Family History of Coronary Artery Disease (Parents, Brothers and Sisters) [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 13473
    No family history | 12307
    Positive family history | 1166
Family History of Cerebrovascular Disease (Parents, Brothers and Sisters) [Count of Participants; unit: Participants] — Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 13468
    No family history | 11960
    Positive family history | 1508
Consumption of Triglyceride (TG) in 3 Month Prior to the Observation Period [Mean (Standard Deviation); unit: Milligram/deciliter (mg/dL)] | 229.2 (101.98)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (Cumulative Incidence) With Specified Cardiovascular Events in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with specified cardiovascular events from start of observation in population of omega-3 fatty acid ethyl esters 2 g user. Specified cardiovascular events were fatal and non-fatal, and defined as major adverse cardiovascular events (cardiovascular death [including sudden death, fatal myocardial infarction, fatal cardiac failure, fatal stroke {cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage} and other cardiovascular death], non-fatal myocardial infarction, and non-fatal stroke [cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage]), angina pectoris requiring coronary revascularization (i.e., percutaneous transluminal coronary angioplasty [PCI] or coronary artery bypass grafting [CABG]), peripheral arterial disease requiring surgery or peripheral arterial intervention.
Time Frame: Up to 36 months
Population: Participants in efficacy analysis set who received both interventions and standard antihyperlipidemic therapy as part of routine medical care. The efficacy analysis set was defined as all participants who completed the survey.
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.5
  12 months | 1.1
  18 months | 1.4
  24 months | 1.9
  30 months | 2.2
  36 months | 2.5

2. Primary Outcome: Percentage of Participants (Cumulative Incidence) With Specified Cardiovascular in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with specified cardiovascular events from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user. Specified cardiovascular events were fatal and non-fatal, and defined as major adverse cardiovascular events (cardiovascular death [including sudden death, fatal myocardial infarction, fatal cardiac failure, fatal stroke {cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage} and other cardiovascular death], non-fatal myocardial infarction, and non-fatal stroke [cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage]), angina pectoris requiring coronary revascularization (i.e., percutaneous transluminal coronary angioplasty [PCI] or coronary artery bypass grafting [CABG]), peripheral arterial disease requiring surgery or peripheral arterial intervention.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.6
  12 months | 1.2
  18 months | 1.6
  24 months | 1.9
  30 months | 2.4
  36 months | 2.7

3. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Death From All Causes (Cardiovascular and Non-cardiovascular Deaths) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with death from all causes (cardiovascular and non-cardiovascular deaths) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.4
  18 months | 0.7
  24 months | 0.9
  30 months | 1.1
  36 months | 1.4

4. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Death From All Causes (Cardiovascular and Non-cardiovascular Deaths) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with death from all causes (cardiovascular and non-cardiovascular deaths) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.2
  12 months | 0.5
  18 months | 0.7
  24 months | 0.9
  30 months | 1.2
  36 months | 1.4

5. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Major Adverse Cardiovascular Events (MACE) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with major adverse cardiovascular events (MACE) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user. MACE included cardiovascular death (including sudden death, fatal myocardial infarction, fatal cardiac failure, fatal stroke [cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage] and other cardiovascular death), non-fatal myocardial infarction, and non-fatal stroke (cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage).
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.3
  12 months | 0.7
  18 months | 0.9
  24 months | 1.2
  30 months | 1.3
  36 months | 1.5

6. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Major Adverse Cardiovascular Events (MACE) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with major adverse cardiovascular events (MACE) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user. MACE included cardiovascular death (including sudden death, fatal myocardial infarction, fatal cardiac failure, fatal stroke [cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage] and other cardiovascular death), non-fatal myocardial infarction, and non-fatal stroke (cerebral infarction, cerebral hemorrhage, and subarachnoid hemorrhage).
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.2
  12 months | 0.6
  18 months | 0.8
  24 months | 1.0
  30 months | 1.2
  36 months | 1.4

7. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With All Cardiovascular Events From in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with all cardiovascular events from start of observation in population of omega-3 fatty acid ethyl esters 2 g user. All cardiovascular events included MACE, angina pectoris requiring hospitalization, angina pectoris requiring coronary revascularization (i.e., PCI or CABG), cardiac failure requiring hospitalization, transient ischaemic attack requiring hospitalization, peripheral arterial disease requiring hospitalization, peripheral arterial disease requiring surgery or peripheral arterial intervention.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.7
  12 months | 1.4
  18 months | 1.8
  24 months | 2.3
  30 months | 2.7
  36 months | 3.1

8. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With All Cardiovascular Events in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with all cardiovascular events from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user. All cardiovascular events included MACE, angina pectoris requiring hospitalization, angina pectoris requiring coronary revascularization (i.e., PCI or CABG), cardiac failure requiring hospitalization, transient ischaemic attack requiring hospitalization, peripheral arterial disease requiring hospitalization, peripheral arterial disease requiring surgery or peripheral arterial intervention.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.7
  12 months | 1.6
  18 months | 2.1
  24 months | 2.6
  30 months | 3.1
  36 months | 3.6

9. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Cardiovascular Death) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (cardiovascular death) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.3
  18 months | 0.4
  24 months | 0.5
  30 months | 0.5
  36 months | 0.7

10. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Cardiovascular Death) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (cardiovascular death) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.3
  18 months | 0.3
  24 months | 0.4
  30 months | 0.5
  36 months | 0.6

11. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Non-fatal Myocardial Infarction) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (non-fatal myocardial infarction) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.1
  18 months | 0.1
  24 months | 0.3
  30 months | 0.3
  36 months | 0.3

12. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Non-fatal Myocardial Infarction) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (non-fatal myocardial infarction) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Never User of Omega-3- Fatty Acid Ethyl Esters 2 g: Participants received standard antihyperlipidemic therapy without omega-3 fatty acid ethyl esters 2 g as part of routine medical care.
Arm/Group | Never User of Omega-3- Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.1
  18 months | 0.2
  24 months | 0.2
  30 months | 0.2
  36 months | 0.3

13. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Non-fatal Stroke) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (non-fatal stroke) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.2
  12 months | 0.3
  18 months | 0.3
  24 months | 0.4
  30 months | 0.5
  36 months | 0.5

14. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Non-fatal Stroke) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (non-fatal stroke) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.2
  18 months | 0.3
  24 months | 0.3
  30 months | 0.4
  36 months | 0.5

15. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Angina Pectoris Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (angina pectoris requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.3
  12 months | 0.5
  18 months | 0.6
  24 months | 0.8
  30 months | 0.9
  36 months | 1.1

16. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Angina Pectoris Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (angina pectoris requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.3
  12 months | 0.6
  18 months | 0.9
  24 months | 1.0
  30 months | 1.2
  36 months | 1.4

17. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Angina Pectoris Requiring Coronary Revascularization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data waspercentage of participants (cumulative incidence) with individual cardiovascular events (angina pectoris requiring coronary revascularization ) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.2
  12 months | 0.4
  18 months | 0.5
  24 months | 0.7
  30 months | 0.8
  36 months | 0.9

18. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Angina Pectoris Requiring Coronary Revascularization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (angina pectoris requiring coronary revascularization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.3
  12 months | 0.5
  18 months | 0.8
  24 months | 0.9
  30 months | 1.1
  36 months | 1.2

19. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Cardiac Failure Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (cardiac failure requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.1
  18 months | 0.2
  24 months | 0.2
  30 months | 0.4
  36 months | 0.4

20. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Cardiac Failure Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (cardiac failure requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.1
  12 months | 0.3
  18 months | 0.4
  24 months | 0.5
  30 months | 0.6
  36 months | 0.7

21. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Transient Ischaemic Attack Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (transient ischaemic attack requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.0
  18 months | 0.0
  24 months | 0.0
  30 months | 0.1
  36 months | 0.1

22. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Transient Ischaemic Attack Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (transient ischaemic attack requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.0
  18 months | 0.1
  24 months | 0.1
  30 months | 0.1
  36 months | 0.1

23. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Peripheral Arterial Disease Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (peripheral arterial disease requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.0
  18 months | 0.1
  24 months | 0.1
  30 months | 0.1
  36 months | 0.1

24. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Peripheral Arterial Disease Requiring Hospitalization) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (peripheral arterial disease requiring hospitalization) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.1
  18 months | 0.1
  24 months | 0.1
  30 months | 0.2
  36 months | 0.2

25. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Peripheral Arterial Disease Requiring Surgery or Peripheral Arterial Intervention) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (peripheral arterial disease requiring surgery or peripheral arterial intervention) from start of observation in population of omega-3 fatty acid ethyl esters 2 g user.
Time Frame: Up to 36 months fatty
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ever User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 6580
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.0
  18 months | 0.0
  24 months | 0.0
  30 months | 0.1
  36 months | 0.1

26. Secondary Outcome: Percentage of Participants (Cumulative Incidence) With Individual Cardiovascular Events (Peripheral Arterial Disease Requiring Surgery or Peripheral Arterial Intervention) in Population of Omega-3 Fatty Acid Ethyl Esters 2 g Never User
Description: Reported data was percentage of participants (cumulative incidence) with individual cardiovascular events (peripheral arterial disease requiring surgery or peripheral arterial intervention) from start of observation in population of omega-3 fatty acid ethyl esters 2 g never user.
Time Frame: Up to 36 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Never User of Omega-3 Fatty Acid Ethyl Esters 2 g
Number analyzed (Participants) | 7784
Percentage of participants
  Start of observation | 0.0
  6 months | 0.0
  12 months | 0.1
  18 months | 0.1
  24 months | 0.1
  30 months | 0.2
  36 months | 0.2

ADVERSE EVENTS:
Time Frame: Up to 36 months
Description: In this survey, only the data of mortality and cardiovascular side effects with Omega-3 fatty acid ethyl esters 2 g (see Other Adverse Event[AE]s table below) were planned to be collected and report. That is, due to observational study, the other AEs data such as serious AEs, non-cardiovascular AEs were not planned to be collected and reported. Reported data were only mortality and side effects data in the population of treatment with Omega-3 fatty acid ethyl esters 2 g.
Groups:
- Omega-3 Fatty Acid Ethyl Esters 2 g: The usual adult dosage for oral use was 2 g of omega-3 fatty acid ethyl esters administered once daily or twice daily immediately after meals for treatment of hyperlipidemia. Participants received both interventions and standard antihyperlipidemic therapy as part of routine medical care. Reported groups were combined in this section because group assignment (groups with or without intervention of omega-3 fatty acid ethyl esters) was conducted after completion of data collection (collection of Case Report Form) in this observational study and collection of data for each group during this study was not planned on the protocol of this study.
Arm/Group | Omega-3 Fatty Acid Ethyl Esters 2 g
All-Cause Mortality (participants affected / at risk) | 74/5859
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 25/6867
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omega-3 Fatty Acid Ethyl Esters 2 g (N=6867)
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 2
Angina pectoris (Cardiac disorders) | 8
Myocardial infarction (Cardiac disorders) | 1
Sudden death (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02285166/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02285166/SAP_001.pdf